CLINICAL TRIAL: NCT04004039
Title: Sarcopenia Mechanism and Therapeutic
Brief Title: Understanding Loss of Muscle Mass and Function
Acronym: SAMANTHA
Status: Withdrawn | Type: Observational
Why Stopped: Application to a CPP
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM U1046 CNRS UMR 9214, Montpellier University (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0272
Record Dates: First submitted 2019-06-07; First posted 2019-07-01 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Sarcopenia
Keywords: Satellite cells; Therapeutic; Aromatic plants
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcopenia is a loss of muscle mass and function that develops during aging. But sarcopenia is also observed in several other conditions: chronic diseases, cancers, viral infections, renal / respiratory insufficiency, immobility, obesity with low physical activity. This sarcopenia is named secondary sarcopenia to distinguish it from the age-associated primary sarcopenia. During prolonged hospitalizations in intensive care, a significant loss of muscular mass and function is also observed. This acute sarcopenia or Intensive Care Unit-Acquired Weakness (ICU-AW) may persist for several months after discharge from hospital. In addition to the loss of autonomy, the reduction of muscle mass has important metabolic implications, ranging from insulin resistance to modification of myokines production. Sarcopenia greatly increases the morbidity and mortality of patients regardless of its cause. The aim of our project is to identify the molecular mechanisms implicated in sarcopenia from different origin. We will particularly focus our work on the metabolic properties, the proliferation/ differentiation and regeneration capacities of the satellite cells (adult muscle stem cells). These satellite cells will be purified from quadriceps biopsies of human volunteers recruited at CHU Montpellier. These satellite cells will also be used to test the ability of some wild aromatic plants from south of France to improve cell survival and differentiation. This will allow us to identify the molecular mechanisms involved in sarcopenia development and identify potential therapeutic molecules.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing quadriceps muscle biopsy as part of the treatment.
* Patient having given their agreement of conservation within the framework of the care of the biological sample (biopsy and blood sample)

Exclusion Criteria:

* Subject refusing the detection of anti-HIV, anti-hepatitis C antibodies, HBS antigen
* Subject treated with anticoagulant, beta blocker, lipid-lowering agent (statin or fibrate), anti-inflammatory, ACE inhibitors, angiotensin 2 receptor antagonist or corticosteroids, including locally.
* Allergic subject to local anesthetics
* History or presence of psychoactive substance abuse
* History of recent abdominal surgery (less than 3 months)
* Subject deprived of liberty by judicial or administrative decision
* Major subject protected by law
* Inability to understand the nature and purpose of the study and / or communication difficulties with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sarcopenic and non-sarcopenic patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Properties and characterization of satellite cells of healthy subjects compared to satellite cells of subjects with sarcopenia. | 6 years
  Properties and characterization of satellite cells of healthy subjects compared to satellite cells of subjects with sarcopenia, 9 outcomes : Diameter of myotubes in culture, Immune properties, Proliferation: cell growth curve, Differentiation: expression of some proteins specific of myotubes as myogenin and troponin T by Western Blotting, Differentiation: expression of troponin T by microscopy and immunofluorescence, Differentiation: expression of some mRNA coding for specific protein by RTqPCR, Transcriptomic analysis, Mitochondria activity: citrate synthase activity, Mitochondria quantity by Western Blot analysis

SECONDARY OUTCOMES:
Reversal of sarcopenia with chemicals compounds extracted from wild aromatic plants from south of France vs control (not treated cells) | 5 years
  Reversal of sarcopenia with chemicals compounds extracted from wild aromatic plants from south of France vs control, 7 outcomes : Diameter of myotubes in culture, Improvement of cell survival (Viability by FACS in % of cells/ml of cell culture media compared to control), Differentiation: expression of some proteins specific of myotubes as myogenin and troponin T by Western Blotting, Differentiation: expression of troponin T by microscopy and immunofluorescence, Differentiation: expression of some mRNA coding for specific protein by RTqPCR, Mitochondria activity: citrate synthase activity, Mitochondria quantity by Western Blot analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Mercier, Pr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC